CLINICAL TRIAL: NCT01322035
Title: Erythrocyte and Adipocyte G6PD Activity Levels Correlate With Differing Degrees of Dyslipidemia, Insulin Resistance and Obesity
Brief Title: Erythrocyte and Adipocyte G6PD Activity Levels in Obesity
Status: Completed | Type: Observational
Sponsor: University of South Alabama (Other)
Responsible Party: Principal Investigator, William Richards, principal investigator, University of South Alabama
Other Study IDs: 09.0027
Record Dates: First submitted 2010-06-23; First posted 2011-03-24 (Estimated); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples(adipose, omentum and liver biopsies)
Oversight: Data Monitoring Committee: No

SUMMARY:
This study compares the improvement of weight, fasting lipid profile (triglycerides, cholesterol, HDL, and LDL) and diabetes after gastric bypass surgery with an improvement in levels of an enzyme called glucose-6-phosphate dehydrogenase (G6PD).

DETAILED DESCRIPTION:
Same as brief summary

ELIGIBILITY:
Inclusion Criteria:

* Age > 19 years of age and <70 years of age
* HGA1c<6.0%
* fasting blood sugar less than 100mg/dL

Exclusion Criteria:

* Taking antidiabetic medications for other indications

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be morbidly obese and undergo Roux-en-Y Gastric bypass surgery. Both Type 2 diabetic and non-diabetic patients will be accepted into the study.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William O Richards, MD, Principal Investigator — University of South Alabama, Department of Surgery
Locations (2):
- United States (2):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - University of South Alabama, Mobile, Alabama

RESULTS

PARTICIPANT FLOW:
Groups:
- Type 2 Diabetic: morbidly obese type 2 diabetic patients
- Nondiabetic: morbidly obese nondiabetic patients
Period: Overall Study
Arm/Group | Type 2 Diabetic | Nondiabetic
Started | 16 | 11
Completed | 8 | 8
Not Completed | 8 | 3
Not completed — Lost to Follow-up | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 2 Diabetic | Nondiabetic | Total
Number analyzed (Participants) | 16 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.20 (2.52) | 44 (3.40) | 45.6 (2.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 7 | 5 | 12
body mass index [Mean (Standard Deviation); unit: kilograms per meter squared] | 45.61 (2.61) | 47.72 (2.92) | 46.67 (2.77)
cholesterol [Mean (Standard Deviation); unit: mg/dL] | 199.10 (12.23) | 208.70 (11.90) | 203.9 (12.07)
triglycerides [Mean (Standard Deviation); unit: mg/dL] | 283.1 (56.25) | 202.40 (43.61) | 242.75 (49.93)
fasting insulin [Mean (Standard Deviation); unit: mIU/L] | 54.89 (19.55) | 36.49 (12.75) | 45.69 (16.15)
homeostatic model assessment insulin resistent [Mean (Standard Deviation); unit: HOMA-IR score] — The HOMA(IR) is a highly specific tool in measuring insulin resistance in patients in both diagnosis of diabetes and its treatment.
  HOMA IR is calculated from blood fasting insulin concentration (μU/ml) × fasting glucose concentration (mmol/L)/22.5 and must be taken at the same point in time.
  Normal healthy subjects have a HOMA(IR) of 1 while subjects with type 2 diabetes have elevated levels of HOMA IR. Higher levels indicate more insulin resistance and therefore a worse outcome measure.
  HOMA-IR score | 30.51 (11.98) | 8.50 (3.10) | 19.51 (7.54)
hemoglobin A 1 c [Mean (Standard Deviation); unit: percent of HbA1c] | 9.38 (0.62) | 5.52 (0.06) | 7.45 (0.34)
fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 207 (17.69) | 93.08 (2.50) | 150.04 (10.10)

OUTCOME MEASURES:

1. Primary Outcome: Measure Erythrocyte G6PD Levels in Diabetic vs. Non-diabetic Morbidly Obese Patients Undergoing Laparoscopic Gastric Bypass.
Description: G6PD levels will be measured various time intervals. G6PD is the rate limiting enzyme of the pentose phosphate pathway that provides NADPH required for lipid synthesis. G6PD overexpression is implicated in insulin resistance, hyperlipidemia and increases in oxidative stress.
Time Frame: G6PD levels will be measured at the following time intervals: Baseline(prior to gastric bypass surgery), 1 week, 6 weeks, and 12 weeks post surgery.
Measure: Mean (Standard Deviation); unit: nM/min/mg
Groups:
- Diabetic: morbidly obese patients
- Nondiabetic: nondiabetic morbidly obese
Arm/Group | Diabetic | Nondiabetic
Number analyzed (Participants) | 8 | 8
nM/min/mg
  Baseline | 3.12 (5.22) | 0.67 (0.46)
  1 week post surgery | 22 (1.39) | 13 (0.14)
  6 week post surgery | 20 (1.39) | 12 (0.14)
  12 week post surgery | 7.58 (9.81) | 11.72 (14.38)
Statistical Analysis 1: Comparison: Diabetic vs Nondiabetic; Test type: Equivalence — 95% confidence limits from standard deviation of the mean were used as the equivalence; p < 0.05, Wilcoxon (Mann-Whitney); 95% confidence limits from standard deviation

2. Secondary Outcome: Measure Adipocyte G6PD Levels in Diabetic vs. Non-diabetic Morbidly Obese Patients Undergoing Laparoscopic Gastric Bypass.
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: nM/min/mg
Arm/Group | Type 2 Diabetic | Nondiabetic
Number analyzed (Participants) | 16 | 11
nM/min/mg
  Baseline | 3.12 (1.39) | 0.67 (0.14)
  1 week postop | 22.1 (3.5) | 13 (2.8)
  6 weeks | 21.9 (3.2) | 12.5 (2.7)
  12 weeks post surgery | 8 (2) | 4.9 (1.5)

3. Secondary Outcome: Measure Omentum G6PD Levels in Diabetic vs. Non-diabetic Morbidly Obese Patients Undergoing Laparoscopic Gastric Bypass.
Time Frame: time of gastric bypass
Measure: Mean (Standard Error); unit: nM/min/mg
Arm/Group | Type 2 Diabetic | Nondiabetic
Number analyzed (Participants) | 8 | 8
nM/min/mg | 13 (3) | 12 (2)

4. Secondary Outcome: Measure Hepatocyte G6PD Levels in Diabetic vs. Non-diabetic Morbidly Obese Patients Undergoing Laparoscopic Gastric Bypass.
Time Frame: time of gastric bypass
Measure: Mean (Standard Error); unit: nM/min/mg
Arm/Group | Type 2 Diabetic | Nondiabetic
Number analyzed (Participants) | 8 | 8
nM/min/mg | 17 (2) | 11.9 (2.1)

ADVERSE EVENTS:
Time Frame: baseline to 12 months
Groups:
- Type 2 Diabetic; Nondiabetic: no adverse events occurred
Arm/Group | Type 2 Diabetic | Nondiabetic
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 0/16 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No